CLINICAL TRIAL: NCT00055081
Title: The Impact of Family CTI on Homeless Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Judith Samuels, The Nathan Kline Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH067148 (NIH); R01MH067148 (NIH); DSIR 82-SEMS
Record Dates: First submitted 2003-02-19; First posted 2003-02-20 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Mental Health
Keywords: Homeless Persons
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Critical Time Intervention

SUMMARY:
The purpose of this study is to examine how services and housing provided for homeless families affect the mental health and behavior of homeless children over time.

DETAILED DESCRIPTION:
This study is a supplement to a parent study which concentrates on the outcomes of homeless mothers who are provided with services and housing. This study will focus on the effects of housing and services on children, who may be the major beneficiaries of such assistance.

Participants are randomly assigned to either receive services and permanent housing or to remain in a homeless shelter without additional assistance. Children and their parents are interviewed separately 3, 9, and 15 months after study entry. The teachers of participating children are surveyed twice during the study.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the parent study
* Homeless and living at a shelter with mother/maternal guardian at the time of study enrollment

Ages: 18 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2002-07; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Internalizing, externalizing, school outcomes | 18 months post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Samuels, MBA, PhD, Principal Investigator — The Nathan S. Kline Institute for Psychiatric Research
Locations (1):
- The Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York, United States